CLINICAL TRIAL: NCT05728853
Title: Is Bioimpedance Analysis Accurate in Transgender Males?
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Signe Graungaard, MSc Clinical Nutrition, Aalborg University Hospital
Other Study IDs: N-20220054
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Transgenderism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trans gender males: Trans gender males in hormonal therapy
  Interventions: Radiation: Assessment of body composition

INTERVENTIONS:
Radiation: Assessment of body composition — Assessment of body composition using BIA and DXA

SUMMARY:
Accurate fat mass and muscle mass assessment is an informative marker of an individual's health. However, the optimal method for assessing body composition in transgender males remains to be determined. Here, the investigators aim to compare body composition estimates in transgender males by bioimpedance analysis using the reference settings for males and females and by

DETAILED DESCRIPTION:
Gender incongruence is defined as a condition in which the gender with which a person identifies does not align with the gender assigned at birth. According to a recent population survey, 0.55% of the Danish population are gender incongruent, and 0.10% define themselves as transgender. There is an equal distribution between trans men and trans women. The treatments include gender-affirming hormone therapy and gender-affirming surgery. Exogenous treatment with sex steroids such as testosterone plays an important role in the distribution of body fat and lean body mass development, and thus induces masculinization of body composition in transgender males.

Body composition is a highly informative marker of an individual's nutrition-related condition and health. Furthermore, it contributes to the identification, diagnosis, and management of several medical conditions. In obesity, the body composition assessment improves the diagnosis and is useful in the monitoring of treatment response, which is central in the management of obesity-related chronic diseases and sarcopenic obesity. Maintaining muscle mass (MM) is important for longevity and health in humans as there is a natural increase in fat mass (FM) and a decrease in MM with age. This leads to an increased risk of cardiovascular disease, type 2 diabetes, several types of cancer, sarcopenia, and even early mortality. However, weight and BMI do not provide insights into the relative contributions of FM and MM on disease risk.

Body composition measured by bioimpedance analysis (BIA) includes FM and lean body mass estimates. The test is inexpensive, readily reproducible and suitable for outpatient clinic patients. Body fat percentage, measured by BIA, reflects body adiposity and is a superior indicator of obesity compared to BMI. Dual x-ray absorptiometry (DXA) is the gold standard distinguishing fat, lean tissue, and bone mineral, thus providing accurate estimates of bone mineral density, FM, and lean soft tissue/fat-free mass (FFM). The main limitations of DXA are that it is expensive, time-consuming, and exposes the subjects to radiation, which may hinder its use at a large scale. As body composition is more accurately assessed by fat percentage and FFM than BMI, it is relevant to consider which methods are most reliable for assessing body composition in transgender males.

We aim to investigate whether estimates of body composition by BIA in transgender males are significantly affected by the use of binary reference values. Furthermore, we aim to compare the body composition estimated by BIA to DXA scans.

ELIGIBILITY:
Inclusion Criteria:

* Trans gender males in hormonal therapy
* Age ≥ 18 years
* Ability to provide informed consent

Exclusion Criteria:

* Inability to comprehend written consent form or provide informed consent
* BMI > 35
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans gender males
Study Population: Transgender males in hormonal therapy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Body fat percentage | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Signe Graungaard, MSc, Principal Investigator — North Denmark Region
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05728853/Prot_000.pdf